CLINICAL TRIAL: NCT04861441
Title: Comparison of Continue Cryotherapy and Standard Ice Packs for Pain Reduction Following Total Shoulder Arthroplasty
Brief Title: Continuous Cryotherapy in Shoulder Arthroplasty Patients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: House staff unable to follow protocol due to short staffing, turnover, and travel nursing.
Sponsor: D. Patrick Williams (Other)
Collaborators: Lake Erie College of Osteopathic Medicine (Other)
Responsible Party: Sponsor-Investigator, D. Patrick Williams, Assistant Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY20100056
Record Dates: First submitted 2021-04-22; First posted 2021-04-27 (Actual); Last update posted 2023-06-23 (Actual); Status verified 2023-06

CONDITIONS: Pain, Shoulder
MeSH Terms: conditions — Shoulder Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Continuous Cryotherapy (Experimental): Subjects will use continuous cryotherapy post operative for pain control
  Interventions: Device: Aircast Cryo Cuff (Shoulder) and Aircast Cryo Cuff I/C Motorized Cooler
- Icepack (Active Comparator): Subjects will use standard icepacks post operative for pain control
  Interventions: Device: Icepacks

INTERVENTIONS:
Device: Aircast Cryo Cuff (Shoulder) and Aircast Cryo Cuff I/C Motorized Cooler — Patient will wear the continuous cryo cuff for a designated period of time and will record their pain and narcotic use post operatively.
  Arms: Continuous Cryotherapy
Device: Icepacks — Standard of care icepacks will be used postoperatively for designated amount of times and patients will record pain and narcotic use post operatively.
  Arms: Icepack

SUMMARY:
This is a randomized prospective study to test if cooling therapies decrease narcotic pain medication use in patients following total shoulder replacement surgery (total shoulder arthroplasty, TSA). Postoperative standard care involves use of ice packs placed on the surgical site for periods of approximately 20 minutes every 2 hours, but they do not provide consistent temperature and can become uncomfortably cold. Continuous cryotherapy (CC) machines provide flow of continuous cooled water (45-55° F) via a cuff placed on the affected sight for several hours. There are mixed results as to whether CC is more beneficial than standard ice pack therapy. This study will address whether CC decreases pain and narcotic pain medication use compared to ice pack therapy in TSA patients. The investigators will monitor both patient-reported pain scores and actual narcotic use to test the hypothesis that use of CC reduces postoperative pain and the need for narcotic pain medication. The results of this study may help establish parameters for non-pharmacologic intervention to reduce patient reliance on narcotic medications.

DETAILED DESCRIPTION:
Prior to the surgical procedure, the patients will be met by one of the coinvestigators or Dr. Williams in the preoperative holding area. At this time, the patients will be administered a questionnaire about their current pain level using a Visual Analog Scale (VAS) of 0-10, where 0 is no pain and 10 is the worse pain imaginable. The questionnaire will be the same questionnaire used after surgery, so questions referencing ice use will be disregarded for this initial interview. After all questions have been answered, patients will receive an interscalene block by the anesthesiology team prior to being brought to the operative suit. Interscalene block routinely performed prior to shoulder arthroplasty at our institution.

At the conclusion of the surgery, a randomly assigned envelope indicating the arm of the study will be opened. At that time, the indicated therapy (ice pack or CC) will be initiated. Ice packs and CC machines will be available and readily accessible for nursing staff to assist study participants. The CC group will use the following protocol:

The CC will be initiated immediately after surgery, with application of the CC cuff in the OR. Temperature will be set to between 45-55°F. The machine will be worn continuously for the first 72 hours postoperatively. The machine is portable and can be taken with the patients as they move about the hospital/home. After the first 72 hours CC will be used as needed. Patients will be encouraged to use the CC whenever their pain is rated 4-5 on the VAS. Prior to discharge, the patient will be instructed on machine use and the at home protocol. The protocol includes when to wear the machine and how to record CC and narcotic use. Written instructions for the protocol and a diary for recording usage will be provided to the patient. The patients will document the time and duration the machine is in use, along with their pain prior to and after use. The protocol will continue through postoperative day 28. Data collection will end a postoperative day 28, though patients may continue to use the machine longer if they choose.

The standard ice therapy group will use the following protocol:

The standard ice therapy will be initiated immediately post-operatively. While in the hospital, ice will be applied for 20 minutes every 2 hours. Upon discharge, ice pack therapy will be applied for 20 minutes every 2 hours while awake. (Patient do not need to wake up every 2 hours to apply ice at night.) After 72 hours post-operative, patient may apply ice therapy for 20 minutes as needed, in 2 hour time increments. Patients will be encouraged to use the ice whenever their pain is rated 4-5 on the VAS. Prior to discharge, the patient will be instructed about ice pack use and the at home protocol. The protocol includes when to use ice and how to record ice usage and narcotic use. Written instructions for the protocol along with a diary will be provided to the patient. Subjects will document the time and duration the standard ice therapy is in use along with their pain prior to and after usage. This will be continued until postoperative day 28, when data will stop being collected. The patient may continue to use icepacks after postoperative day 28 if they choose.

The postoperative pain regimen will begin in the hospital. Both groups will have scheduled Tylenol, 650 mg every 6 hours. Patients will also receive 3 doses of 15 mg of Toradol starting on postoperative day 1. They will also have oxycodone available, with 5 mg for VAS of 1-3, 10 mg for VAS of 4-6, and 15 mg for VAS of 7-10. If patients do not tolerate oxycodone, or require additional narcotics for pain, these will be adjusted. This adjustment will be offset by using a conversion to morphine equivalents for data analysis purposes. Throughout the hospital stay, narcotic use will be recorded in terms of morphine equivalents by using the Medication Administration Record (MAR) tab within PowerChart.

Subjective VAS pain scores will be obtained by nursing every 4 to 8 hours as this is required for the administration of oxycodone per protocol. Along with having nursing obtain the pain score, one of the co-investigators will conduct postoperative interviews with patients at 24 and 48 hours using the same questionnaire that was used preoperatively with ice use questions included. The same questions will be asked to both groups. As most patients discharge on postoperative day 2, the investigators will defer further interview until postoperative day 7.

Upon discharge, patients will be provided the following pain regimen protocol: Tylenol 650 mg every 6 hours for VAS 1-3, Tylenol 650 mg plus 600 mg Ibuprofen every 6 hours for VAS 4-6, and Tylenol 650 mg plus 5 mg Oxycodone every 6 hours. Prior to the patient taking medication, they will asked to record the following information on provided diary: current VAS score, pain medication taken, and therapy usage (either cryo or ice packs).

On postoperative day 7, a phone interview will be conducted to again evaluate the patient's pain and document narcotic use during the first postoperative week. For patient's pain score, the investigators will ask what they felt was their average score throughout the week. For the narcotic use the investigators will ask them how many pills they have taken while at home. Conversion will be used to standardize all values to morphine equivalents. Ice pack or CC machine usage will be reviewed and documented. Medication and ice use will also be recorded on the patient diary to monitor consistency of responses.

An in-person interview using the same format as phone interviews will occur at their postoperative visit approximately 14 days after surgery. This is the standard follow-up appointment for patients. Patients will turn in their written logs and narcotic use will be monitored by counting the remaining pills in the patient's prescription bottle. At this time, another diary sheet will be provided for the patient along with a prepaid envelope to OSME.

A second phone interview will occur on postoperative day 28, when the investigators anticipate ice have ceased. Pain scores, narcotic use, and the date(s) of cessation, if applicable, will be recorded. At this time, patients will be instructed to mail in their diaries using the prepaid envelope. Patient can continue using the respective therapy as needed at this point. If patients are still taking narcotics at day 28 postoperatively, this will be noted, and the investigators will continue to help control their pain.

ELIGIBILITY:
Inclusion Criteria:

* Patients between the age of 55 and 80 who are indicated for a TSA, including both anatomic (maintaining anatomic location of the ball and socket in the shoulder) and reverse (reverses where the ball and socked are placed) total shoulder arthroplasties.

Exclusion Criteria:

* Patients undergoing:

  * revision total shoulder arthroplasty
  * TSA for a fracture
* Patients with a history of narcotic abuse.
* Patients unwilling or unable to receive and interscalene block
* Patients with Raynaud's disease, vasospastic disease, or other circulatory dysfunction
* Patients with cold hypersensitivity, decreased skin sensitivity related to temperature
* Patients with central ports, PICC lines, or other indwelling IV access on the affected side.

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-10-22 (Actual); Primary Completion 2022-06-24 (Actual); Study Completion 2022-06-24 (Actual)

PRIMARY OUTCOMES:
Continuous monitoring of pain control | Up to post operative day 28
  Pain control will be self reported using a visual analog scale (VAS) for pain. The scale will be from 1 to 10 with 1 being being less severe pain and 10 being more severe pain
Continuous monitoring of narcotic use | Up to post operative day 28
  Subjects will record narcotic post operatively and this will be converted to morphine equivalents.

CONTACTS AND LOCATIONS:
Overall Officials: D. Patrick Williams, DO, Principal Investigator — UPMC Hamot, Department of Orthopaedics
Locations (1):
- UPMC Hamot, Erie, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No